CLINICAL TRIAL: NCT00815152
Title: Coping With High Grade Glioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI transferred to new institution.
Sponsor: Duke University (Other)
Collaborators: National Brain Tumor Foundation(NBTF) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00012826; NCT00849498 (obsolete NCT alias)
Record Dates: First submitted 2008-12-26; First posted 2008-12-29 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2010-10

CONDITIONS: Glioma
Keywords: high grade glioma; Coping skills intervention; caregivers
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Twenty five caregivers will randomly be assigned to receive active coping skills training and 25 caregivers will randomly receive usual care at The Preston Robert Tisch Brain Tumor Center at Duke.
  Interventions: Behavioral: coping skills intervention training
- 2 (Placebo Comparator): Caregivers that will receive ususal care.
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: coping skills intervention training — The strategies will include ways to improve problem solving, communication skills, and managing activities.
  Arms: 1
Behavioral: usual care — The ususal care at the Preston Robert Tisch Brain Tumor Center
  Arms: 2

SUMMARY:
1. Purpose and Objective:

   To determine the feasibility and short- and long-term efficacy of an empirically-based CST intervention (Keefe et al.) with caregivers of patients with primary malignant brain cancer.
2. Study Activities and Population Group:

   The target sample will be 20 caregiver-patient dyads. Using a randomized controlled, prospective design, potentially eligible participants will be identified at the time of initial consultation (see Figure 1). Outcomes will be assessed at baseline, post-intervention (3 months post-randomization), 6 months post-randomization, and every 4 months up to 2-years in the event that the patient dies.
3. Data Analysis and Risk/Safety Issues:

With only 10 subjects per group we do not have statistical power for direct hypothesis testing. Nevertheless, p-values will be presented for some analyses (chi-square tests, t-tests, and Spearman correlations) simply to aid in interpretation of results. In no way will these p-values be used to declare statistical significance or non-significance of the test results. Accordingly, the primary focus will be the means, variances, and covariances of the study endpoints, as well as the change scores in these endpoints across the study intervention and their 95% confidence limits.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility and short- and long-term efficacy of an empirically-based CST intervention (Keefe et al.) with caregivers of patients with primary malignant brain cancer. The target sample will be 20 caregiver-patient dyads. The caregiver may be a spouse/partner, family member or friend,. Additional inclusion criteria will include: (1) caregiver provides a weekly minimum of 4 hours of caregiving; (2) caregiver is 18 years or older; (3) caregiver reading level at or above 8th grade; (4) caregiver sufficiently fluent in English; (5) the patient shows evidence of problems in depression, fatigue, sleep disturbance, and/or cognitive impairment as per the treating neuro-oncologist; (6) the caregiver and patient are willing to be randomized to treatment or usual care condition; (7) patient is within 3 months of initial diagnosis; (8) patient has life expectancy of at least 6 months or more; (9) the caregiver is willing to participate in treatment sessions using a telephone. If a patient dies during the active 12-week study phase, then the caregiver will be transitioned to the follow-up phase or removed from the study and, if needed, be referred for appropriate psychiatric or psychological treatment.

Using a randomized controlled, prospective design, potentially eligible participants will be identified at the time of initial consultation. Outcomes will be assessed at baseline, post-intervention (3 months post-randomization), 6 months post-randomization, and every 4 months up to 2-years in the event that the patient dies. If the subject is assigned to the intervention, they will be asked to complete 12 weeks of a coping skills training intervention. The coping skills intervention will consist of six telephone conversations during which they will learn strategies to reduce stress. The strategies will include ways to improve problem solving, communication skills, and managing activities. The subject will also be asked to complete a packet of questionnaires which will take about 1 hour to do. The subject will be asked to complete the questionnaires multiple times during the study (before the coping skills intervention, during the week after the coping skills intervention, and 3 months after the coping skills intervention). If the subject is assigned to the usual care condition, they will be asked to complete assessments at the same time intervals as caregivers in the active coping skills intervention. In either condition, in the event that the patient dies, the caregiver will also be asked to complete assessments every four months for one year. Patients will be asked to participate in sessions and complete questionnaires as they are able to.

ELIGIBILITY:
Inclusion Criteria:

The caregiver may be a spouse/partner, family member or friend. Additional inclusion criteria will include:

1. caregiver provides a weekly minimum of 4 hours of caregiving;
2. caregiver is 18 years or older;
3. caregiver reading level at or above 8th grade;
4. caregiver sufficiently fluent in English;
5. the patient shows evidence of problems in depression, fatigue, sleep disturbance, and/or cognitive impairment as per the treating neuro-oncologist;
6. the caregiver and patient are willing to be randomized to treatment or usual care condition;
7. patient is within 3 months of initial diagnosis;
8. patient has life expectancy of at least 6 months or more;
9. the caregiver is willing to participate in treatment sessions using a telephone. If a patient dies during the active 12-week study phase, then the caregiver will be transitioned to the follow-up phase or removed from the study and, if needed, be referred for appropriate psychiatric or psychological treatment.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To explore the effects of a coping skills training (CST) intervention on distress, self-efficacy and other related outcomes among caregivers of high grade glioma patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bart Brigidi, PhD, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States